CLINICAL TRIAL: NCT01063361
Title: Effect of Low Glycemic Index Diets (With Pulses) on Glucose Control in Non-Insulin Dependent Diabetics
Brief Title: Low Glycemic Index Diets (With Pulses) in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Saskatchewan Pulse Growers (Other); Pulse Canada (Other)
Responsible Party: Principal Investigator, David Jenkins, Principle Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-192
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pulse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low glycemic Index Diet (Experimental): Low glycemic Index Diet, emphasizing pulses
  Interventions: Dietary Supplement: Low glycemic index diet with pulses
- High Cereal Fibre Diet (Active Comparator)
  Interventions: Dietary Supplement: High Cereal Fibre

INTERVENTIONS:
Dietary Supplement: Low glycemic index diet with pulses — Subjects will be advised to follow a diabetic diet, using low glycemic index foods, emphasizing pulses.
  Arms: Low glycemic Index Diet
Dietary Supplement: High Cereal Fibre — Subjects will be advised to follow a healthy high fibre diabetic diet.
  Arms: High Cereal Fibre Diet

SUMMARY:
Healthy individuals with type 2 diabetes will receive intensive counseling on food selection to improve glucose control using either high cereal fiber dietary strategies or low glycemic index foods emphasizing dried legumes and their products. The treatments will last 3 months with bloods taken for HbA1c, glucose and blood lipids. If the study shows a benefit for either or both diets, then use of high fiber and/or low glycemic index foods in the diet may provide another potential way to improve glucose control and lower cholesterol levels in non-insulin dependent diabetes.

ELIGIBILITY:
Inclusion Criteria: Men and women with type 2 diabetes who

* are treated with oral hypoglycemic agents at a stable dose for at least 8 weeks
* have a HbA1c in the range of 6.5% to 8.5% at screening and at the visit prior to randomization
* have diabetes diagnosed >6 months
* have maintained stable weight for 2 months (within 3%)
* have a valid OHIP card and a family physician
* if prescribed lipid medication, have taken a stable dose for at least 2 weeks
* if prescribed blood pressure medication, have taken a stable dose for at least 1 week
* can keep written food records, with the use of a digital scale

Exclusion Criteria: Individuals who

* take insulin
* take steroids
* have GI disease (gastroparesis, celiac disease, ulcerative colitis, Crohn's Disease, IBS)
* have had a major cardiovascular event (stroke or myocardial infarction) in the past 6 months
* take warfarin (Coumadin)
* have had major surgery in the past 6 months
* have a major debilitating disorder
* have clinically significant liver disease (AST or ALT > 130 U/L), excluding NAFL or NASH
* have hepatitis B or C
* have renal failure (high creatinine > 150 mmol/L)
* have serum triglycerides ≥ 6.0 mmol/L
* have a history of cancer, except non-melanoma skin cancer (basal cell, squamous cell)
* have food allergies to study food components
* have elevated blood pressure (> 145/90) unless approved by GP
* have acute or chronic infections (bacterial or viral)
* have chronic inflammatory diseases (e.g. rheumatoid arthritis, lupus; ulcerative colitis)
* have other conditions which in the opinion of any of the investigators would make them unsuitable for the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
change in HbA1c | from prestudy and week 0, to end of treatment weeks 8, 10, and 12
serum lipids | from prestudy and week 0, to end of treatment weeks 8, 10, and 12

SECONDARY OUTCOMES:
fasting glucose | from prestudy and week 0, to end of treatment weeks 8, 10, and 12
change in weight, waist and hip circumference | weeks 0, 12
blood pressure | from prestudy and week 0, to end of treatment weeks 8, 10, and 12
creatine, urea, and c-peptides in 24 hour urine collection | 0, 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jenkins DJ, Kendall CW, Augustin LS, Mitchell S, Sahye-Pudaruth S, Blanco Mejia S, Chiavaroli L, Mirrahimi A, Ireland C, Bashyam B, Vidgen E, de Souza RJ, Sievenpiper JL, Coveney J, Leiter LA, Josse RG. Effect of legumes as part of a low glycemic index diet on glycemic control and cardiovascular risk factors in type 2 diabetes mellitus: a randomized controlled trial. Arch Intern Med. 2012 Nov 26;172(21):1653-60. doi: 10.1001/2013.jamainternmed.70. PMID 23089999